CLINICAL TRIAL: NCT01570010
Title: The Norwegian Dietary Guidelines and Colorectal Cancer Survival Study
Brief Title: Effect of Norwegian Food Based Dietary Guidelines on Chronic Diseases in CRC Survivors
Acronym: CRC-NORDIET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); Finnish Institute for Health and Welfare (Other Government); University Hospital, Akershus (Other); Norwegian Cancer Society (Other); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Rune Blomhoff, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CRC-NORDIET study; 2011/836 (Other: REK Sør-Øst)
Record Dates: First submitted 2012-03-22; First posted 2012-04-04 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group (n = 250) receives an intensive dietary intervention lasting for 12 months and a subsequent maintenance intervention for 14 years. Both groups are offered equal general advice of physical activity.
  Interventions: Other: Norwegian food based dietary guidelines
- Control group (Other): The control group (n = 250) receives no dietary intervention other than standard clinical care. Both groups are offered equal general advice of physical activity.
  Interventions: Other: Norwegian food based dietary guidelines

INTERVENTIONS:
Other: Norwegian food based dietary guidelines — several means will be applied to guide participarts to cohere to the dietary guidelines including access to clinical nutritionists, free food, food discounts, cooking courses, cookbook/recipies, study website, organized physical activity, etc
  Other Names: Typisk norsk

SUMMARY:
The current study is designed to gain a better understanding of the role of a healthy diet aimed at dampening inflammation and oxidative stress on long-term disease outcomes and survival in colorectal cancer patients. Since previous research on the role of diet for colorectal cancer survivors is limited, the study may be of great importance for this cancer population.

DETAILED DESCRIPTION:
Men and women aged 50-80 years diagnosed with primary invasive colorectal cancer (Stage I-III) are invited to this randomized controlled, parallel two-arm trial 2-9 months after curative surgery. The intervention group (n = 250) receives an intensive dietary intervention lasting for 12 months and a subsequent maintenance intervention for 14 years. The control group (n = 250) receives no dietary intervention other than standard clinical care. Both groups are offered equal general advice of physical activity. Patients are followed-up at 6 months and 1, 3, 5, 7, 10 and 15 years after baseline. The study center is located at the Department of Nutrition, University of Oslo, and patients are recruited from two hospitals within the South-Eastern Norway Regional Health Authority. Primary outcomes are disease-free survival and overall survival. Secondary outcomes are time to recurrence, cardiovascular disease-free survival, compliance to the dietary recommendations and the effects of the intervention on new comorbidities, intermediate biomarkers, nutrition status, physical activity, physical function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer (ICD10 C18-20) TNM Stage I-III

Exclusion Criteria:

* TNM stage 0 or IV

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5, 10 and 15 years
  Disease-free survival (DFS) (events are defined as detection of local recurrence or metastasis or any second cancer or death from any cause)
Overall survival | 10, 15 years
  Overall survival (OS) (event is defined as death from any cause)

SECONDARY OUTCOMES:
Time to recurrence | up to 15 years
  Events are defined as detection of local recurrence or metastasis
CVD -free survival | up to 15 years
  Events of CVD (ICD-10; chapter I) or death from any cause
CRC-specific survival | up to 15 years
  death due to CRC
Total cancer-specific survival | up to 15 years
  death due to CRC or any other cancer
Inflammatory disease-specific survival | up to 15 years
  death due to inflammatory disease
Cardiovascular (CVD)-specific survival | up to 15 years
  death due to CVD
New morbidity of other diet-related chronic diseases | up to 15 years
  e.g. ischemic coronary heart disease, cerebrovascular disease, thromboembolic disease, type 2 diabetes, obesity, hypertension and chronic obstructive pulmonary disease
Dietary intake and nutritional status | up to 15 years
  Questionnaires, food records, clinical consultation
Physical activity and function | up to 15 years
  Questionnaires, arm band, physical tests
Nutrition biomarkers | up to 15 years
  e.g., carotenoids, fatty acids, 25-hydroxy vitamin D etc
Body composition | up to 15 years
  DXA, CT, BIA
Anthropometric measures | up to 15 years
  eg weight, waist and hip circumference
Biomarkers for inflammation and oxidative stress | up to 15 years
  e.g. isoprostanes, cytokines
Transcription- and epigenetic profiles | up to 15 years
  sequencing and arrays
Biomarkers for cardiovascular disease, metabolic syndrome, type 2-diabetes, thromboembolic disease and cancer | up to 15 years
  e.g. blood pressure, total/LDLcholesterol, HbA1c, CRP, IL-6, IL-10, TNFα
Health related quality of life and fatigue | up to 15 years
  Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Rune Blomhoff, Professor, Principal Investigator — University of Oslo
Locations (3):
- Norway (3):
  - Akershus University Hospital, Lørenskog
  - University of Oslo, Oslo
  - Oslo University Hospital, Oslo

REFERENCES:
- [Result] Henriksen HB, Raeder H, Bohn SK, Paur I, Kvaerner AS, Billington SA, Eriksen MT, Wiedsvang G, Erlund I, Faerden A, Veierod MB, Zucknick M, Smeland S, Blomhoff R. The Norwegian dietary guidelines and colorectal cancer survival (CRC-NORDIET) study: a food-based multicentre randomized controlled trial. BMC Cancer. 2017 Jan 30;17(1):83. doi: 10.1186/s12885-017-3072-4. PMID 28137255
- [Result] Henriksen C, Paur I, Pedersen A, Kvaerner AS, Raeder H, Henriksen HB, Bohn SK, Wiedswang G, Blomhoff R. Agreement between GLIM and PG-SGA for diagnosis of malnutrition depends on the screening tool used in GLIM. Clin Nutr. 2022 Feb;41(2):329-336. doi: 10.1016/j.clnu.2021.12.024. Epub 2021 Dec 18. PMID 34999327
- [Result] Alavi DH, Henriksen HB, Lauritzen PM, Kvaerner AS, Sakinis T, Langleite TM, Henriksen C, Bohn SK, Paur I, Wiedswang G, Smeland S, Blomhoff R. Quantification of adipose tissues by Dual-Energy X-Ray Absorptiometry and Computed Tomography in colorectal cancer patients. Clin Nutr ESPEN. 2021 Jun;43:360-368. doi: 10.1016/j.clnesp.2021.03.022. Epub 2021 Apr 15. PMID 34024541
- [Result] Henriksen HB, Berntsen S, Paur I, Zucknick M, Skjetne AJ, Bohn SK, Henriksen C, Smeland S, Carlsen MH, Blomhoff R. Validation of two short questionnaires assessing physical activity in colorectal cancer patients. BMC Sports Sci Med Rehabil. 2018 May 29;10:8. doi: 10.1186/s13102-018-0096-2. eCollection 2018. PMID 29854408
- [Result] Henriksen HB, Carlsen MH, Paur I, Berntsen S, Bohn SK, Skjetne AJ, Kvaerner AS, Henriksen C, Andersen LF, Smeland S, Blomhoff R. Relative validity of a short food frequency questionnaire assessing adherence to the Norwegian dietary guidelines among colorectal cancer patients. Food Nutr Res. 2018 Feb 22;62. doi: 10.29219/fnr.v62.1306. eCollection 2018. PMID 29545734
- [Derived] Eklo RR, Alavi DT, Konglevoll DM, Kolle A, Henriksen HB, Rising R, Blomhoff R, Olsen T. Predictive equations commonly used in clinics underestimate resting energy expenditure compared with whole-room indirect calorimetry in colorectal cancer survivors. Am J Clin Nutr. 2026 Jan 27:101209. doi: 10.1016/j.ajcnut.2026.101209. Online ahead of print. PMID 41611086
- [Derived] Henriksen HB, Kolle A, Stenling A, Paur I, Bohn SK, Broto P, Tronstad TS, Blomhoff R, Berntsen S. Spillover effect of a dietary intervention on physical activity in a randomized controlled trial with colorectal cancer patients. Int J Behav Nutr Phys Act. 2025 May 9;22(1):54. doi: 10.1186/s12966-025-01757-0. PMID 40346639
- [Derived] Nordengen AL, Krutto A, Kvaerner AS, Alavi DT, Henriksen HB, Kolle A, Henriksen C, Smeland S, Bohn SK, Zheng C, Shaposhnikov S, Collins AR, Blomhoff R. Plant-based diet and oxidative stress-induced DNA damage in post-surgery colorectal cancer patients: Results from a randomized controlled trial. Free Radic Biol Med. 2025 Jun;233:240-249. doi: 10.1016/j.freeradbiomed.2025.03.047. Epub 2025 Apr 1. PMID 40180023
- [Derived] Alavi DT, Henriksen HB, Lauritzen PM, Zucknick M, Bohn SK, Henriksen C, Paur I, Smeland S, Blomhoff R. Effect of a one-year personalized intensive dietary intervention on body composition in colorectal cancer patients: Results from a randomized controlled trial. Clin Nutr ESPEN. 2023 Oct;57:414-422. doi: 10.1016/j.clnesp.2023.06.037. Epub 2023 Jul 11. PMID 37739688